CLINICAL TRIAL: NCT06260956
Title: Expecting Mother's Study of Consumption or Avoidance of Peanut and Egg
Acronym: ESCAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Kirsi Jarvinen-Seppo, Chief of Pediatric Allergy and Immunology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U01-ROC-001; 1U01AI173032 (NIH)
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Allergy and Immunology; Peanut and Nut Allergy; Egg Allergy; Food Allergy in Infants; Food Allergy Peanut
MeSH Terms: conditions — Hypersensitivity; Nut and Peanut Hypersensitivity; Egg Hypersensitivity; Peanut Hypersensitivity | interventions — Economics; SAV4 protein, Arabidopsis

STUDY DESIGN:
Intervention Model Description: National, parallel, two arm (one-to-one allocation), single blinded, randomized controlled trial.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, the subjects must know which arm they are assigned to, however, biostatistician and investigators will be blinded to study assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Consumption (Active Comparator): Subjects must consume peanuts and peanut products and egg and egg products.
  Interventions: Behavioral: Consumption
- Arm 2 Avoidance (Active Comparator): Subjects must avoid eating peanuts and peanut products and egg and egg products.
  Interventions: Behavioral: Avoidance

INTERVENTIONS:
Behavioral: Consumption — Subjects consume peanut and egg from 27 weeks of pregnancy through the first 4 months feeding breastmilk to their infant.
  Arms: Arm 1 Consumption
Behavioral: Avoidance — Subjects avoid eating peanut and egg from 27 weeks of pregnancy through the first 4 months feeding breastmilk to their infant.
  Arms: Arm 2 Avoidance

SUMMARY:
Peanut allergy is the most common cause of fatal and near-fatal food-allergic reactions and egg allergy is among the two most common causes of food-induced anaphylaxis. The proposed research will explore the development of sensitization to these food(s) in infants based on maternal consumption or avoidance during pregnancy and breastfeeding.

DETAILED DESCRIPTION:
The goals of this study include defining the role of egg and peanut consumption or avoidance during pregnancy and via human milk in food sensitization and identifying the underlying biological mechanisms leading to sensitization or tolerance. The study population will include 500 mother/infant dyads who plan to exclusively feed breastmilk to healthy infants. We expect approximately 25% will be recruited locally and the rest from across the United States. This is a national, parallel, two arm, one-to-one allocation, single blinded, randomized controlled trial. Each arm of the study defines maternal diet from 27 weeks gestation through their baby's fourth month with some consuming peanut and egg and some avoiding these foods.

ELIGIBILITY:
Inclusion Criteria:

• o Subject must be able to understand and provide informed consent.

* English-speaking adults, 18 years or older. (Spanish speaking adults may be included after consent document is translated and Spanish speaking study representatives are available to conduct and answer questions during informed consent process and for study follow up.)
* Maternal consent must be provided for infants.
* Pregnant women from the time pregnancy is confirmed until 27 weeks of gestation.
* Self-reported at time of enrollment:

  * no chronic inflammatory conditions that require long-term systemic immunosuppressive medications in first or second trimester
  * carrying a fetus with a first-degree relative (i.e., mother, father, full sibling) with any self-reported or physician-diagnosed allergic disease (asthma, allergic rhinitis, atopic dermatitis, or food allergy).
* Intend to give their infant their own breast milk for more than 3 months.
* Can confidently say they have eaten PN and egg and have tolerated consumption with no food allergy reactions.
* Willing to be randomized to consumption or avoidance diet.
* Uncomplicated pregnancy (no gestational diabetes, no preeclampsia, no hyperemesis gravidarum), self-reported at time of enrollment.

Exclusion Criteria:

* Inability or unwillingness of subject to give written informed consent or comply with study protocol.
* Known history of renal/liver/cardiac insufficiency in the mother or infant.
* Pregnant women with PN or egg allergy.
* Pregnant women who refuse to eat PN (or peanut products) and/or eggs.
* Physician diagnosed immunodeficiency in the mother or infant.
* Current, diagnosed, mental illness or current, diagnosed, or self-reported, drug or alcohol abuse that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements.
* Past or current medical problems or findings from medical history that are not listed above, which, in the opinion of the investigator, may pose additional risks to the mother or infant from participation in the study, may interfere with the subject's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To understand the mechanisms whereby maternal diet either positively or negatively affects the development of their infant from the womb through the first few months of life, it is necessary to recruit healthy pregnant women.
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Egg or peanut sensitization | four months
  Determine the proportion of high-risk infants who have developed egg or peanut sensitization at four months (prior to introduction of these foods to the infant).

SECONDARY OUTCOMES:
Peanut and egg specific IgG and IgG4 | four months
  Levels of infant peanut and egg specific IgG and IgG4
Antibodies in maternal blood | four months
  Quantify egg- and PN-specific IgG and IgG4 antibody concentrations in maternal blood measured during pregnancy and at four months.
Egg allergy | 12 months
  Questionnaire for parents to report any signs of egg allergy in their child.
Egg and peanut specific IgE | four months
  Measure levels of infant egg- and peanut-specific IgE.

OTHER OUTCOMES:
Exploratory: Peanut sensitization | four months
  The proportion of high-risk infants who have developed peanut sensitization
Exploratory: Egg sensitization | four months
  Proportion of infants who develop egg sensitization.
Exploratory: Symptoms | four months
  Questionnaire for parents to report symptoms of non-IgE mediated food allergy
Exploratory: Peanut sensitization 12 months | 12 months
  Questionnaire for parents to report signs of peanut allergy
Mechanistic: antigen level | four months
  Measure PN and egg antigen levels in house dust and human milk
Mechanistic: IgG levels | four months
  Quantify PN- and egg-specific IgG antibody levels in maternal serum and human milk.
Mechanistic: T cell | four months
  Phenotype infant T cell populations in cord blood and infant blood.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Per NIH policy